CLINICAL TRIAL: NCT04647006
Title: Comparison of Transoral Endoscopic Thyroidectomy Vestibular Approach and Open Conventional Thyroidectomy for Inflammatory Responses, Pain and Patient Satisfaction: A Prospective Study
Brief Title: Comparison of TOETVA and Conventional Thyroidectomy
Acronym: TOETVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MUnlu (Other Government)
Collaborators: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Sponsor-Investigator, MUnlu, Principal Investigator, Başakşehir Çam & Sakura City Hospital
Organization: Başakşehir Çam & Sakura City Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mehmet Taner Unlu
Record Dates: First submitted 2020-10-06; First posted 2020-11-30 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Thyroid; Thyroid Nodule; Surgery
Keywords: thyroidectomy; transoral; TOETVA
MeSH Terms: conditions — Thyroid Diseases; Thyroid Nodule | interventions — Thyroid (USP)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Thyroidectomy (Other): Conventional Thyroidectomy
  Interventions: Procedure: thyroid
- Transoral endoscopic thyroidectomy vestibular approach (Active Comparator): Transoral endoscopic thyroidectomy vestibular approach
  Interventions: Procedure: thyroid

INTERVENTIONS:
Procedure: thyroid — Conventional Thyroidectomy and Transoral endoscopic thyroidectomy vestibular approach

SUMMARY:
Introduction-Objective:

The application of transoral endoscopic thyroidectomy vestibular approach (TOETVA) is gradually increasing recently. However, it is not clear whether TOETVA is a true minimally invasive thyroidectomy compared to open conventional thyroidectomy.

In this study, we aimed to evaluate the TOETVA and open conventional thyroidectomy techniques in terms of postoperative inflammatory response, pain and patient satisfaction.

Material and Method:

In this prospective study, 40 female patients between the ages of 18-65 were divided into 2 groups of 20 patients: TOETVA: 20 patients, open thyroidectomy: 20 patients. Operation time, inflammatory response with IL-6, white blood cell (WBC) and C-reactive protein (CRP), postoperative pain, postoperative complications and patient satisfaction were evaluated in both groups.

DETAILED DESCRIPTION:
The application of transoral endoscopic thyroidectomy vestibular approach (TOETVA) is gradually increasing recently. However, it is not clear whether TOETVA is a true minimally invasive thyroidectomy compared to open conventional thyroidectomy.

In this study, we aimed to evaluate the TOETVA and open conventional thyroidectomy techniques in terms of postoperative inflammatory response, pain and patient satisfaction.

This non-randomized prospective clinical study was performed in our clinic between September 2019 and January 2020 with the approval of the Sisli Hamidiye Etfal Training and Research Hospital Ethics Committee (Ethics committee date: 19/03/2019, number: 2313).

In the study, it was planned to form 2 groups with 20 patients in each, performing conventional open thyroidectomy (OTG) (Group 1) or transoral endoscopic thyroidectomy vestibular approach (TOETVA) (TTG) (Group 2). All patients who agreed to participate in the study were informed about both surgical techniques and complications, and their written consent was obtained. Patients took part in Group 1 or Group 2 according to their own preferences.

During this study, 43 patients underwent thyroidectomy. Patients who did not comply with the study criteria were excluded from the study. 43 female patients were selected from these patients who were eligible for the study. Of these patients, 3 patients who were converted to open surgery in the TTG group were excluded from the study, and a total of 40 patients were included in the study.

All surgeries were performed by an experienced endocrine surgeon.

Conventional thyroidectomy: After neck extension with a thyroid pillow and patient positioning, thyroidectomy and/or central neck dissection was performed using a 4 to 6cm collar transverse incision. Subplatysmal flap dissection was applied up to the sternal notch inferiorly and to the thyroid cartilage superiorly, and through the mid line of the strap muscles, the thyroid gland was reached. After receiving a vagus nerve impulse, upper pole dissection was performed under the guidance of IONM. Identification and monitoring of recurrent laryngeal nerves (RLNs) and external branch of the superior laryngeal nerves (EBSLNs) were carried out systematically.

TOETVA: All patients received preoperative chlorhexidine mouthwash and preoperative intravenous amoxicillin/clavulanic acid was administered for prophylaxis. Orotracheal intubation was performed. A slight extension posture was given to the neck with a pillow placed under the shoulder, and the patients were placed in 15 degrees of Trendelenburg position. Skin and oral cavity were wiped with povidone iodine. A central 1.5-2 cm transverse incision was performed in the middle of the distance between the first vermillion inner edge and the inferior labial frenulum in the oral vestibule. Through the peripheral fibers of the submucosa and orbicularis oris muscle, the jaw tip was reached with a monopolar electrocautery between the two mentalis muscles deep in the subdermal layer. From this incision, 50 cc of 1/500000 adrenaline-saline solution was applied to the anterior neck with a Veress needle. A surgical field was created from this incision by dissection of thyroid cartilage with Kelly forceps. The surgical field was formed by blunt dissection from the incision in the subplatysmal area, up to both sternocleidomastoid muscles (SCMs) leading edge and to the sternal notch in the inferiorly with the blunt type tunnel probe. For the 30° camera from the central incision, 10 mm blunt tipped port was entered and operation was performed under 6 mmHg CO 2 pressure and 15 L/min CO 2 flow rate. In addition, with 3-4 silk sutures placed on the front neck, the skin is mechanically hung and an optimal working area is provided. A vertical 5 mm incision was made from the lateral side of the canine tooth and edge of vermillion at both sides, and two working channels were created parallel to the 10 mm port. Subplatysmal workspace was opened completely with Hook cautery and Harmonic scalpel. Strap muscles were opened in midline, and dissected over thyroid gland. The strap muscles were retracted by a transcutaneous 2/0 silk suture. Thyroid isthmus is divided. The upper pole was dissected, controlled with the EBSLN monitoring probe, and the thyroid vessels were separated from the thyroid capsule with Ultracision. The superior parathyroids are identified and dissected and protected. The recurrent laryngeal nerve was viewed at the entrance of the larynx and introduced towards proximally. The Berry region was separated close to the thyroid capsule to protect RLN. Inferior parathyroids have been identified and protected. The thyroid gland was separated from the trachea. The thyroid gland was placed in the endobag placed through the 10 mm port and extracted. The same surgical procedures were applied to the opposite lobe in total thyroidectomy. Following bleeding control, RLN (R2) and vagus (V2) signals were measured with IONM probe and recorded. Surgicel was placed into the surgical field. The midline was closed with 3/0 polyglactin sutures. No drain was used in any patient. Intraoral incisions were sutured with 4/0 polyglactin. 24-hour pressure dressing was applied to the chin.

The upper pole vessels were separated on the thyroid capsule with bipolar cautery. In lateral dissection of the thyroid lobe, RLN was identified in the region where it crosses with the inferior thyroid artery (ITA). Then, RLN was fully dissected up to its entry through the larynx under the cricopharyngeal muscle (CP muscle). Preserving parathyroids, ITA branches were separated from the capsule. R2 and V2 signals were measured after bleeding control. Surgicel® was placed in the surgical field and strap muscles were reapproximated with 3/0 polyglactin. The subcutaneous tissue was sutured separately with polyglactin. The skin was reapproximated subcutaneously with polyglactin.

Inflammatory Response: Preoperative, postoperative 2nd hour, 1st day and 2nd day CRP (C-reactive protein), WBC (White blood cell), IL-6 (Interleukin 6) levels were measured to evaluate the inflammatory response in all patients. To measure IL-6, blood samples were collected from patients, centrifuged, then stored at -80oC. After all the serum were collected, they were evaluated using the Human IL-6 ELISA kit. To evaluate postoperative hypoparathyroidism, postoperative first day calcium, phosphorus and parathormone values were checked. Hypocalcemic patients were controlled weekly and evaluated clinically and with laboratory values.

Postoperative pain and analgesia: As a standard in terms of pain palliation, all patients received 4*1 500 mg paracetamol intravenously and 3*1 100 mg tramadol HCl on the first day; 3*1 500 mg paracetamol intravenously on the second day in the postoperative period.

Pain intensity of the patients was evaluated with the Visual Analogue Scale (VAS) score (0 to 10) on the 2nd and 12th hour, 1st and 2nd days postoperatively. Lower lip, lower chin and anterior neck area pain were evaluated separately with VAS score. VAS scores were determined by patients by marking the intensity of pain on the ruler, which was marked as 0 for the absence of pain and as 10 for the most severe pain sensation.

Patient satisfaction was evaluated on postoperative 15th and 30th days in both groups. Patients were asked to evaluate and score the operation in general and in terms of cosmesis (1: bad and 4: very good). In addition, the patients were asked which surgery (TOETVA or conventional thyroidectomy) they would prefer if they would have the operation again.

Vocal cord examination with fiberoptic laryngoscopy was performed to all patients in the preoperative period and within the first 2 days postoperatively by an independent otorhinolaryngologist. Control examinations were planned for patients with vocal cord paralysis at the 15th day, 1st, 2nd, 4th and 6th months postoperatively.

Intraoperative and postoperative complications of patients were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Must be aged 18 to 65 years
* Benign thyroid disease, with FNAB results Bethesda 3,4 or below 1 cm + Bethesda V, VI
* Thyroid volume less than 50 cm3
* Largest nodule diameter must be less than 4 cm
* No previous neck, chin and oral surgery
* No vocal cord paralysis for any reason
* In the preoperative period, clinically euthyroid and laboratory results in the euthyroid state
* Agreed to participate in the study were included in the study..

Exclusion Criteria:

* Patients with a FNAB result of Bethesda V, VI over 1 cm,
* Planning of central and/or lateral neck dissection due to thyroid cancer
* Patients with thyroid volume greater than 50 cm3
* Secondary intervention cases
* Patients with accompanying hyperparathyroidism
* Patients with preoperative vocal cord paralysis (VCP)
* Patients with ASA score III and IV
* Patients who were started with TOETVA and converted to the conventional method intraoperatively

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2020-01-28 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Evaluate the TOETVA and Open Conventional Thyroidectomy Techniques in Terms of Postoperative Inflammatory Response by CRP (C-reactive protein) | 4 days
  To evaluate the TOETVA and open conventional thyroidectomy techniques in terms of postoperative inflammatory response; CRP (C-reactive protein) levels were measured in all patients for evaluating the inflammatory response at preoperative, postoperative second hour, first day and second day.
Evaluate the TOETVA and Open Conventional Thyroidectomy Techniques in Terms of Postoperative Inflammatory Response by WBC (white blood cells) | 4 days
  To evaluate the TOETVA and open conventional thyroidectomy techniques in terms of postoperative inflammatory response; WBC (white blood cells) levels were measured in all patients for evaluating the inflammatory response at preoperative, postoperative second hour, first day and second day.
Evaluate the TOETVA and Open Conventional Thyroidectomy Techniques in Terms of Postoperative Inflammatory Response by IL-6 (Interleukin 6) | 4 days
  To evaluate the TOETVA and open conventional thyroidectomy techniques in terms of postoperative inflammatory response; IL-6 (Interleukin 6) levels were measured in all patients for evaluating the inflammatory response at preoperative, postoperative second hour, first day and second day.
Evaluate the Postoperative Pain after TOETVA and Open Conventional Thyroidectomy Techniques Assessed by the Visual Analogue Scale | 4 days
  Pain intensity of the patients was evaluated with the Visual Analogue Scale (VAS) score (0 to 10) on the 2nd and 12th hour, 1st and 2nd days postoperatively. Lower lip, lower chin and anterior neck area pain were evaluated separately with VAS score. VAS scores were determined by patients by marking the intensity of pain on the ruler, which was marked as 0 for the absence of pain and as 10 for the most severe pain sensation.
Comparison of Postoperative Patient Satisfaction Between Conventional Thyroidectomy and TOETVA | 1 month
  Patient satisfaction was evaluated on postoperative 15th and 30th days in both groups. Patients were asked to evaluate and score the operation in general and in terms of cosmesis (1: bad and 4: very good). In addition, the patients were asked which surgery (TOETVA or conventional thyroidectomy) they would prefer if they would have the operation again.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Uludag, 1, Study Director — Sisli Hamidiye Etfal Research Hospital
Locations (1):
- Sisli Etfal Research Hospiatl, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No